CLINICAL TRIAL: NCT02543476
Title: SUPREME-HN A Retrospective Cohort Study of PD-L1 in Recurrent and Metastatic Squamous Cell Carcinoma of Head and Neck (SCCHN)
Acronym: SUPREME-HN
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4193R00002
Record Dates: First submitted 2015-08-25; First posted 2015-09-07 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: PD-L1 status, biomarkers, prevalence, SCCHN, overall survival
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Archival tumor tissues samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients' group with tumor sample: SCCHN patients having available archived tumor sample(s).

SUMMARY:
This is a retrospective international, multi-center, non-interventional cohort study based on use of data derived from established medical records and secondary analysis of archival tumor samples. The study will collect data on patient and tumor characteristics, PD-L1 status, patterns of treatment, and clinical outcomes, in up to 600 adult patients with recurrent/metastatic SCCHN. SCCHN of interest for this study are defined as the diseases falling into specific ICD-10 or International Classification of Diseases, Ninth Revision (ICD-9) codes (Table 1), depending on anatomical sub-site of the primary tumor.

For patient selection, the date of diagnosis of recurrent/metastatic disease will be used as the index date. The patient selection period extends from the 1st March 2011 to the 30th June 2015. This allows for the inclusion of patients with tumor samples of approximately ≤ 5 years age, and ensures approximately 10 months follow-up for living patients recruited at last day of the enrollment window. All patients with a diagnosis of recurrent/metastatic SCC of the oral cavity (tongue, gum, floor of mouth, and other/unspecified part of the mouth), oropharynx, hypopharynx, or larynx during that period will be considered for inclusion in the study (Figure 1). Patients will be identified and followed up through their medical records until death or end of data collection in approximately 20 centers in the US, Asia and Europe.

Patients' demographic, clinical characteristics, and medical history will be described. Clinical outcomes including PFS, best response, duration of response, and ORR will be described for the first line and second line of therapy (if any), and OS will be collected A mandatory archived tumor samples will be used to determine PD-L1 status. If a patient has more than one suitable tissue sample, the most recent sample will be used as the mandatory tissue sample. Where available, additional tumor samples obtained at any other time points of the disease will be also collected (optional).

The enrolment target is up to 600 patients. Statistical analyses will be performed for the whole cohort, per PD-L1 status and for predefined subgroups.

DETAILED DESCRIPTION:
Background/Rationale:

Programmed cell death protein 1 (PD-1) is an immune inhibitory receptor that interacts with two ligands, programmed death ligand 1 (PD-L1) and ligand 2 (PD-L2). PD-1 pathway is a major immune checkpoint which has been implicated in adaptive immune resistance of squamous cell carcinoma of the head and neck (SCCHN) tumors, particularly in those associated with human papillomavirus (HPV) infection. Based on an internal analysis performed by AstraZeneca (AZ), it is reported that approximately 25% of cases of SCCHN express PD-L1. Tumoral PD-L1 expression status correlates closely with response to anti-PD-1/anti PD-L1 antibodies Durvalumab (MEDI4736) is an immunoglobulin G1 kappa monoclonal antibody with high affinity and selectivity for PD-L1 and no binding to PD-L2, which is in development for the treatment of patients with recurrent or metastatic SCCHN.

This non-interventional study (NIS) aims to generate and provide data on the prognostic value of PD-L1 status in patients with recurrent/metastatic SCCHN.

Objectives and Hypotheses:

Primary objective:

To determine the prognostic value of PD-L1 status in terms of overall survival (OS) in patients with recurrent/metastatic SCCHN. Overall survival after diagnosis of recurrent/metastatic SCCHN will be assessed in PD-L1 positive and PD-L1 negative patients and in predefined sub-groups (e.g., HPV status, HIV status, smoking history, heavy alcohol use, anatomical sub-site of primary tumor, and prior exposure to radiation therapy).

Secondary objectives:

Secondary objectives are to perform the following in a) all patients meeting the eligibility criteria, b) all patients per availability of tumor sample (not available, available at any setting), and c) all patients with available tumor sample at any time, at the time of first line therapy, or at the second line therapy per PD-L1 status (positive, negative, unknown/not done):

1. To describe the relevant demographic and clinical characteristics of patients, stratified by PD-L1 status
2. To describe first line treatment choices, and where available, subsequent treatment choices
3. To describe investigator-assessed tumor response for first line and second line of therapy (if any), including: best response, duration of response where applicable, and objective response rate (ORR)
4. To describe investigator-assessed progression-free survival (PFS) for first line and second line of therapy (if any).

Exploratory objectives:

1. To perform additional biomarker research on tumor samples (depending on tissue availability and volume).
2. If feasible, to assess agreement of PD-L1 status in samples obtained at different time points (e.g., before and after chemotherapy or radiation therapy).

Methods:

Study design:

This is a retrospective international, multi-center, non-interventional cohort study based on use of data derived from established medical records and secondary analysis of archival tumor samples. The study will collect data on patient and tumor characteristics, PD-L1 status, patterns of treatment, and clinical outcomes, in up to 600 adult patients with recurrent/metastatic SCCHN.

For patient selection, the date of diagnosis of recurrent/metastatic disease will be used as the index date. The patient selection period extends from the 1st March 2011 to the 30th June 2015. This allows the inclusion of patients with tumor samples of approximately ≤ 5 years age, and ensures approximately 10 months follow-up for living patients recruited at last day of the enrolment window. All patients with a diagnosis of recurrent/metastatic squamous cell carcinoma (SCC) of oral cavity (tongue, gum, floor of mouth, and other/unspecified part of the mouth), oropharynx, hypopharynx, or larynx during that period will be considered for inclusion in the study. Patients will be identified and followed up through their medical records until death or end of data collection (approximately Q4 2016).

Patients' demographic and clinical characteristics, and medical history will be described. Clinical outcomes including PFS, best response, duration of response, and ORR will be described for the first and second lines of therapy(if any), and OS will be collected. A mandatory archived tumor sample will be used to determine PD-L1 status. If a patient has more than one suitable tissue sample, the most recent sample will be used as the mandatory tissue sample. Where available, additional tumor samples obtained at any other time points of the disease will be also collected (optional).

Statistical analyses will be performed for the whole cohort, per PD-L1 status and for predefined subgroups.

Data Source(s):

The study will be implemented in a total of approximately 20 sites in the US, Asia and Europe. Data will be abstracted from patient's hospital medical records until death, or end of data collection. Archival tumor samples will be retrieved and tested by immunohistochemistry to assess the PD-L1 status of the tumor. Where there is sufficient tissue quantity, the expression of other biomarkers will also be evaluated.

Study Population:

Unselected patient population representative of patients who may receive MEDI4736 in the real life setting.

Exposure(s): The primary variable is the PD-L1 status (positive or negative) in the overall patient population. Archived tissue samples, including samples from the primary site, lymph nodes or distant metastatic sites, will be used to determine PD-L1 status. PD-L1 status will be determined by immunohistochemistry (IHC) using a validated assay.

Outcome(s):

Overall survival will be assessed. Additionally, the following clinical outcomes will be described for first line and second line treatments for recurrent and/or metastatic disease: investigator-assessed best tumor response, duration of response where applicable, and investigator-assessed PFS. ORR (sum of complete and partial responses) will be derived from investigator-assessed best responses and described for first line and second line therapies (if any).

Patient characteristics, disease characteristics, and patterns of treatment will be captured and described.

Sample Size Estimation:

The primary objective of this study is to estimate the prognostic value of PD-L1 status in terms of OS in patients with recurrent/metastatic SCCHN. The available sample size is not known a priori and will be driven by the number of patients at selected sites with available tissue. However, assuming that PD-L1 status distribution is approximately 25% positive and 75% negative status, that the median OS in these patients is 10 months, that the study will accrue uniformly over 52 months with 10 months follow-up from the last patient entering and that survival times are exponentially distributed, the illustrations of hazard ratios it would be possible to detect with 80% power (2-sided alpha 0.05) over various sample sizes are given in the table below.

HR to detect Number of deaths Number of patients (Total) 0.3 30 40 0.4 51 68 0.5 74 112 0.6 136 196 0.7 278 396 HR: Hazard ratio These illustrations do not take account of the fact that the binary prognostic factor of interest (PD-L1 status) may be correlated with other covariates and hence could over-estimate the power of the various sample sizes (Bernardo et al, 2000). The sample size (number of events) required when no correlation is assumed should be multiplied by 1/(1-R2) to account for an R2 > 0 (Hsieh and Lavori, 2000). The correlation is not currently known. Additionally, a proportion of patients will not have PD-L1 status available. Given these uncertainties, a sample size of up to 600 patients is felt to be adequate.

Statistical Analysis:

Descriptive analyses on patient characteristics, treatment choices and treatment outcomes will be conducted.

Time to event data (OS, PFS) including rates of affected patients will be assessed described using the Kaplan-Meier method. Two-sided 95% CIs will be provided for the main statistical estimators.

OS and PD-L1 status will be described in subgroups, including but not limited to the following:

* Per anatomical sub-site of primary tumor
* Per HPV status
* Per HIV status
* Per smoking history
* Per alcohol consumption history
* Per prior exposure to radiation therapy
* Per types of treatment regimens
* By performance status at diagnosis of recurrent/metastatic disease. The prognostic value of PD-L1 status will be investigated using a Cox proportional hazards model. Additional covariates to be included in the model will be described in the statistical analysis plan.

ELIGIBILITY:
Inclusion criteria:

1. Provision of subject informed consent (or consent from next of kin/legal representative if applicable) for use of the data and retrieval of tumor sample, according to local regulations 2. Adult patient (≥ 18 years old) 3. Patient with histologically confirmed SCCHN of oral cavity (tongue, gum, floor of mouth, other/unspecified part of the mouth), oropharynx, hypopharynx or larynx 4. Patient with recurrent or metastatic SCCHN diagnosed between 01 March 2011 and 30 June 2015 5. Mandatory archival tissue sample (most recent) from the primary site, a lymph node or a distant metastatic site:

* Tissue sample less than 5 years old (compared to date of retrieval) if provided as complete block (preferred option) or as section cut within 60 days of shipment from site prior to testing 6. Optional archival tissue samples taken at other time points of the disease from the primary site, a lymph node or a distant metastatic site (where available):
* Tissue sample less than 5 years old (compared to date of retrieval) if provided as complete block (preferred option) or as section cut within 60 days of shipment from site prior to testing.

Exclusion criterion:

1. Treatment for SCCHN with anti-CTLA-4, anti-PD-1, anti-PD-L1, or anti-PD-L2 antibodies, or any other antibody with known immunomodulatory effect.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have progressed on or after first line platinum-based chemotherapy regimen for recurrent/metastatic SCCHN and started second line therapy for recurrent/metastatic SCCHN between the 1st January 2010 and the 31st December 2014. Two parallel patient cohorts will be recruited for this study: patients with available tumor sample for determination of PD-L1 status at first and/or second line setting (independently of actual PD-L1 results), and patients without available tumor sample.
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

PRIMARY OUTCOMES:
Prognosis of PD-L1 positive status in the patient population with available tumor sample | From diagnosis to index day, expected to be up to 36 months
  PD-L1 status: positive-negative status measured on tumor slides. Positivity corresponds to more than 25% of tumor cells with membrane positivity for PD-L1. The primary objective of this study is to estimate the prognostic value of PD-L1 status in terms of OS in patients with recurrent/metastatic SCCHN

SECONDARY OUTCOMES:
Exposure to risk factors - alcohol (e.g. Number of participants with alcohol consumption and amount of consumption per day) | At index date, approximately +/- 2 months
  As recorded in the files. Measure of alcohol consumption in number of alcohol units per day. Patients will be categorized based on amount of consumption
Exposure to risk factors - tobacco (e.g. Number of participants with current or past tobacco consumption and amount of consumption per day) | At index date, approximately +/- 2 months
  As recorded in the files. Patients will be categorized according to smoking status at the index date and where available tobacco consumption in Pack years will be obtained from the files as recorded
Exposure to risk factors - Human Immunodeficiency Virus (e.g. Number of participants positive for Human Immunodeficiency Virus) | At index date, approximately +/- 2 months
  Positive/negative to Human Immunodeficiency Virus
Exposure to risk factors - Human papillomavirus (e.g. Number of participants positive for Human papillomavirus) | At index date, approximately +/- 2 months
  Positive/negative to Human papillomavirus
Disease characteristics - performance status WHO criteria | At index date approximately +/- 2 months
  Ranging from 0 to 4 (0: fully active; 4: completely disabled)
Disease characteristics -performance status Karnofsky criteria | At index date approximately +/- 2 months
  Ranging from 20 to 100 with increment of 10 (100: normal, 20: very sick, hospital admission necessary)
Disease characteristics -performance status ECOG criteria | At index date approximately +/- 2 months
  Ranging from 0 to 4 (0: fully active; 4: completely disabled)
Lines of therapy description (e.g. Treatment lines patterns per participants' population) | From First line therapy to end of data collection, expected to be up to 120 months
  Number of therapy lines and duration per patient: will be calculated based on start and stop dates of therapy. Treatment regimen will also be recorded
Clinical outcomes -Best response to treatment line | From First line therapy to end of data collection, expected to be up to 100 months
  The best response of patients whose cancer shrinks or disappears after treatment (as recorded, range from complete response to progression.)
Clinical outcomes - Survival rate | From index date to end of data collection, expected to be up to 85 months
  Time between index date and death/end of participation to study
Complications (from second line therapy for recurrent/metastatic SCCHN) | Complications (from second line therapy for recurrent/metastatic SCCHN) During or shortly after second line therapy, expected to be up to 3 months
  Characterization of most current complications related to treatment (from an existing list)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Pai, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital; Ezra Cohen, M.D., Principal Investigator — University of California San Diego Moores Cancer Center
Locations (18):
- United States (9):
  - Research Site, La Jolla, California
  - Research Site, Atlanta, Georgia
  - Research Site, Hyattsville, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Charlotte, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
- Research Site, Leipzig, Saxony, Germany
- Research Site, Athens, Greece
- Italy (2):
  - Research Site, Legnago (VR), Verona
  - Research Site, Milan
- Japan (2):
  - Research Site, Osaka, Osaka
  - Research Site, Kōtoku, Tokyo-To
- Research Site, Seoul, South Korea
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Seville

REFERENCES:
- [Derived] Pai SI, Cohen EEW, Lin D, Fountzilas G, Kim ES, Mehlhorn H, Baste N, Clayburgh D, Lipworth L, Resteghini C, Shara N, Fujii T, Zhang J, Stokes M, Wang H, Twumasi-Ankrah P, Wildsmith S, Khaliq A, Melillo G, Shire N. SUPREME-HN: a retrospective biomarker study assessing the prognostic value of PD-L1 expression in patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck. J Transl Med. 2019 Dec 26;17(1):429. doi: 10.1186/s12967-019-02182-1. PMID 31878938
- See also: D4193R00002_CSRSynopsisFINAL_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3948&filename=D4193R00002_CSRSynopsisFINAL_Redacted.pdf